CLINICAL TRIAL: NCT06120647
Title: Molecular Mechanisms Underpinning Sarcopenic Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Responsible Party: Principal Investigator, William Apro, Associate Professor, The Swedish School of Sport and Health Sciences
Other Study IDs: 2019-04016
Record Dates: First submitted 2023-10-10; First posted 2023-11-07 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Sarcopenic Obesity; Obesity; Sarcopenia; Aging
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Amino Acids, Essential

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skeletal muscle biopsies from m. vastus lateralis and venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sarcopenic obesity: Age: 70-80 years Men, ALM/W < 25.7 %, body fat % > 35 Women, ALM/W < 19.7 %, body fat % > 40
  Interventions: Dietary Supplement: Essential amino acids (EAA)
- Non-sarcopenic obese: Age: 70-80 years Men, ALM/W > 25.7 %, body fat % > 35 Women, ALM/W > 19.7 %, body fat % > 40
  Interventions: Dietary Supplement: Essential amino acids (EAA)
- Non-sarcopenic lean: Age: 70-80 years Men, ALM > 7.0 kg/m2, body fat % < 25 Women, ALM > 5.5 kg/m2, body fat % < 32
  Interventions: Dietary Supplement: Essential amino acids (EAA)
- Young lean: Age: 18-40 years Men, ALM > 7.0 kg/m2, body fat % < 25 Women, ALM > 5.5 kg/m2, body fat % < 32
  Interventions: Dietary Supplement: Essential amino acids (EAA)

INTERVENTIONS:
Dietary Supplement: Essential amino acids (EAA) — intake of 240 mg EAA per kg lean body mass after a resistance exercise session

SUMMARY:
The coexistence of obesity and sarcopenia results in sarcopenic obesity, a high-risk geriatric condition associated with metabolic perturbations and several co-morbidities. Despite the rising numbers of older adults diagnosed with sarcopenic obesity, few studies have characterized this condition on the muscle cell and systemic level. This study sought to comprehensively assess the influence of sarcopenic obesity on muscle and blood-related parameters and compare it to non-sarocopenic obese and non-sarcopenic lean older adults.

ELIGIBILITY:
Inclusion Criteria:

* Body fat % in accordance with previously defined criteria
* Free of smoking (since 10 years)
* Able to walk without assistance
* Able to perform bilateral leg extension exercise

Exclusion Criteria:

* History of or present disease of myocardial, vascular, endocrine, hepatic, renal, pulmonary or neuromuscular origin
* Uncontrolled hypo/hypertension
* Use of anticoagulants (Warfarin, Trombyl)
* Use of metformin or other anti-diabetic medications
* Poor appetite and unexplained weight loss (4,5 kg) over the past 6 months
* Active malignancy
* Present infection
* Dementia or delirium
* Other conditions that may interfere with the study protocol in the opinion of the PI

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The elderly participants will be community-dwelling living in the greater Stockholm metropolitan area. Participants will be recruited through local senior clubs, online communities, advertisement and word of mouth.
  The young participants will be living in the greater Stockholm metropolitan area. Participants will be recruited through university forums, online communities, advertisement and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Fiber type-specific cell signalling | 1 hour after ingestion of essential amino acids and resistance exercise
  This measure will be investigated during an experimental trial in which the participants are subjected to an acute bout of resistance exercise followed by the ingestion of essential amino acids (240 mg/kg lean mass). During this 3 hour time period, the participants will donate two muscle biopsies, one before exercise and the second one 1 hour after exercise. Cell signalling networks related to muscle mass regulation will be examined in these biopsy samples. The signal will be measured using Western blotting and the signal obtained is expressed in relation to baseline (adjusted volume intensity).

SECONDARY OUTCOMES:
Skeletal muscle fiber characteristics | 1 hour prior to ingestion of essential amino acids and resistance exercise
  Fiber type-specific area measured using immunofluorescence microscope in muscle biopsies collected at baseline (prior to ingestion of essential amino acids and resistance exercise). Unit of measurement is square micrometers (µm^2).
Whole body muscle volume | 1 hour
  Indices of muscle volume and fat infiltration obtained with magnetic resonance imaging (MRI). Unit of measurement is cubic centrimeters (cm^3).
Whole body glucose tolerance | 2 hours
  Oral glucose tolerance test in which the participants will ingest a standardized glucose drink and blood glucose levels will be monitored throughout a period of 2 hours. Unit of measurement is mmol/L glucose.
Accelerometer-assessed physical activity levels | 1 week
  Hip-worn accelerometer data (Actigraph GT3X) collected over 7 consecutive days. Unit of measurement is steps per day.
Isometric and isokinetic leg muscle strength | 1 hour
  Muscle performance will be evaluated at a single timepoint during the study using IsoMed2000 dynamometer. Participants will perform a maximal isometric contraction at 60 degrees of knee flexion. Unit of measurement is Newton meter (N-m).

CONTACTS AND LOCATIONS:
Overall Officials: William Apró, PhD, Principal Investigator — The Swedish School of Sport and Health Sciences and Karolinska Institute, Stockholm Sweden
Locations (1):
- The Swedish School of Sport and Health Sciences, Stockholm, Sweden

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT06120647/SAP_000.pdf